CLINICAL TRIAL: NCT03952130
Title: A Prospective, Randomized, Double-Blind Comparison of LY900014 to Insulin Lispro in Combination With Insulin Glargine or Insulin Degludec in Adults With Type 1 Diabetes
Brief Title: A Study of LY900014 Compared to Insulin Lispro (Humalog) in Adults With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16829; I8B-FH-ITSD (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro; Insulin Glargine; insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY900014 (Experimental): Participants received 100 units per milliliter (U/mL) LY900014 subcutaneously (SC) 0-2 minutes before each meal with either basal insulin glargine or insulin degludec given SC once daily.
  Interventions: Drug: LY900014; Drug: Insulin Glargine; Drug: Insulin Degludec
- Insulin Lispro (Humalog) (Active Comparator): Participants received 100 U/mL insulin lispro SC 0-2 minutes before each meal with either basal insulin glargine or insulin degludec given SC once daily.
  Interventions: Drug: Insulin Lispro; Drug: Insulin Glargine; Drug: Insulin Degludec

INTERVENTIONS:
Drug: LY900014 — Administered SC
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014
Drug: Insulin Lispro — Administered SC
  Other Names: LY275585; Humalog
  Arms: Insulin Lispro (Humalog)
Drug: Insulin Glargine — Administered SC
Drug: Insulin Degludec — Administered SC

SUMMARY:
The purpose of this study is to see if LY900014 compared to insulin lispro (Humalog), both in combination with insulin glargine or insulin degludec, is safe and effective in participants with type 1 diabetes (T1D).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have T1D for at least 1 year prior to screening and continuously using insulin for at least 1 year.
* Participants must have HbA1c of ≥7.0 and ≤10.0%.
* Participants must have been treated for at least 90 days prior to screening with either multiple daily injection(s) (MDI) or premixed analog/human insulin regimens at least twice daily.
* Participants must have body mass index (BMI) of ≤35.0 kilograms per square meter (kg/m2).

Exclusion Criteria:

* Participants must not have used other anti-hyperglycemic medications or therapies (inhaled, oral or injectable) except for metformin within 90-days prior to screening.
* Participants must not have had more than 1 severe hypoglycemic episode within 6 months prior to screening.
* Participants must not have had more than 1 hospitalization related to hyperglycemia or diabetic ketoacidosis within 6 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (30):
- Argentina (3):
  - Centro de Investigaciones Metabólicas (CINME), CABA, Buenos Aires
  - Centro Médico Viamonte, CABA, Buenos Aires
  - Cent Priva Especiali Médicas Ambulatorias Inve Clin CEMAIC, Córdoba
- China (24):
  - The Second People's Hospital of Hefei, Hefei, Anhui
  - Dongguan people's hospital, Dongguan, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Shantou University Medical College No.2 Affiliated Hospital, Shantou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang, Henan
  - The First People's Hospital of Changde City, Changde, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First Hospital of Nanjing, Nanjing, Jiangsu
  - Sir Run Run Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - No.2 Hospital Affiliated to Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Jiangsu Province Hospital, Nanjing, Nanjing
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Beijing Peking Union Medical College Hospital, Beijing
  - Shanghai Putuo District Center Hospital, Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai
- Mexico (3):
  - Unidad de Investigaci�n Cl�nica Cardiometabolica de Occidente, Guadalajara, Jalisco
  - Unidad de patologia Clinica, Guadalajara, Jalisco
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, N.L.

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of LY900014 Compared to Insulin Lispro (Humalog) in Adults With Type 1 Diabetes — https://www.lillytrialguide.com/en-US/studies/type-1-diabetes/ITSD#?postal=

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Lispro (Humalog): Participants received 100 units per milliliter (U/mL) insulin lispro subcutaneously (SC) 0-2 minutes before each meal with either basal insulin glargine or insulin degludec given SC once daily.
- LY900014: Participants received 100 U/mL LY900014 SC 0-2 minutes before each meal with either basal insulin glargine or insulin degludec given SC once daily.
Period: Overall Study
Arm/Group | Insulin Lispro (Humalog) | LY900014
Started | 178 | 176
Received at Least One Dose of Study Drug | 178 | 176
Completed | 176 | 170
Not Completed | 2 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 5

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Lispro (Humalog) | LY900014 | Total
Number analyzed (Participants) | 178 | 176 | 354
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.60 (13.84) | 40.30 (13.42) | 42.00 (13.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 82 | 160
  Male | 100 | 94 | 194
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 141 | 144 | 285
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 31 | 27 | 58
  More than one race | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 21 | 18 | 39
  China | 141 | 144 | 285
  Mexico | 16 | 14 | 30
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. It is measured to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 7.82 (0.91) | 7.87 (0.95) | 7.85 (0.93)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A. It is measured to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) mean was determined by mixed model repeated measures (MMRM) model with Baseline + Pooled Country + Number of Bolus at Study Entry Stratum + Type of Basal at Lead-in Stratum + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and at least one post-baseline HbA1c data.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 165 | 161
Percentage of HbA1c | -0.28 (0.063) | -0.21 (0.064)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; Test type: Non-Inferiority — Noninferiority margin = 0.4% for HbA1c; LS Mean Difference = 0.07, 95% CI 2-sided [-0.11 to 0.24]

2. Secondary Outcome: 1-hour Postprandial Glucose (PPG) Excursion During Mixed-Meal Tolerance Test (MMTT)
Description: A standardized MMTT was used to characterize postprandial glucose control following administration of the study insulin. Serum glucose measured at 1-hour timepoint after the start of meal minus fasting serum glucose. LS mean was determined by analysis of covariance (ANCOVA) model with Baseline + Pooled Country + Hemoglobin A1c Stratum at Baseline + Use of Metformin at Study Entry + Type of Basal at Lead-in Stratum + Treatment (Type III sum of squares) as variables.
Time Frame: Week 26
Population: All randomized participants with baseline and at least one post-baseline 1-hour PPG excursion data.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 141 | 147
milligrams per deciliter (mg/dL) | 102.8 (4.23) | 85.0 (4.14)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; Test type: Superiority; p = 0.003, ANCOVA; LS Mean Difference = -17.8, 95% CI 2-sided [-29.4 to -6.1]

3. Secondary Outcome: 2-hour PPG Excursion During MMTT
Description: A standardized MMTT was used to characterize postprandial glucose control following administration of the study insulin. Serum glucose measured at 2-hour timepoint after the start of meal minus fasting serum glucose. LS mean was determined by analysis of covariance (ANCOVA) model with Baseline + Pooled Country + Hemoglobin A1c Stratum at Baseline + Use of Metformin at Study Entry + Type of Basal at Lead-in Stratum + Treatment (Type III sum of squares) as variables.
Time Frame: Week 26
Population: All randomized participants with baseline and at least one post-baseline 2-hour PPG excursion data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 140 | 147
mg/dL | 142.2 (5.63) | 116.7 (5.49)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; Test type: Superiority; p = 0.001, ANCOVA; LS Mean Difference = -25.5, 95% CI 2-sided [-41.1 to -10.0]

4. Secondary Outcome: Rate of Severe Hypoglycemia
Description: Severe hypoglycemia is defined as an event requiring assistance of another person to administer carbohydrate, glucagon, or other resuscitative actions. Rate of severe hypoglycemia events per 100 years during a defined period was calculated by total number of severe hypoglycemia episodes within the period divided by the cumulative days on treatment from all participants within that treatment group *36525 days.
Time Frame: Baseline through Week 26
Population: All randomized participants who received at least one dose of study drug and had baseline, at least one post-baseline hypoglycemic data.
Measure: Number; unit: Events per 100 participant years
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 177 | 176
Events per 100 participant years | 6.88 | 5.87
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; Test type: Other; p = 0.834, Empirical method; Relative rate = 0.85, 95% CI 2-sided [0.19 to 3.77]

5. Secondary Outcome: Rate of Documented Symptomatic Post Meal Hypoglycemia
Description: Documented symptomatic post meal hypoglycemia is an event during which typical symptoms of hypoglycemia are accompanied by blood glucose (BG) of ≤70 mg/dL [3.9 millimole per liter (mmol/L)]. The rate of documented symptomatic post meal hypoglycemia per year during a defined period is calculated by the total number of documented symptomatic post meal hypoglycemia events within the period divided by the cumulative days on treatment from all participants within that treatment group *365.25.
Time Frame: Baseline through Week 26
Population: as for outcome 4
Measure: Number; unit: Events per participant per year
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 177 | 176
Events per participant per year
  <=30 minutes post meal | 0.11 | 0.09
  <=1 hour post meal | 0.75 | 1.20
  <=2 hours post meal | 3.80 | 4.52
  <=4 hours post meal | 10.2 | 12.4
  >1 to <=2 hours post meal | 3.05 | 3.32
  >2 to <=4 hours post meal | 6.40 | 7.87
  >4 hours post meal | 14.2 | 10.5
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; <=30 minutes post meal; Test type: Other; p = 0.983, Negative binomial regression; Relative rate = 1.00, 95% CI 2-sided [0.72 to 1.38]
Statistical Analysis 2: Comparison: Insulin Lispro (Humalog) vs LY900014; <=1 hour post meal; Test type: Other; p = 0.076, Negative binomial regression; Relative rate = 1.61, 95% CI 2-sided [0.95 to 2.74]
Statistical Analysis 3: Comparison: Insulin Lispro (Humalog) vs LY900014; <=2 hours post meal; Test type: Other; p = 0.409, Negative binomial regression; Relative rate = 1.19, 95% CI 2-sided [0.79 to 1.79]
Statistical Analysis 4: Comparison: Insulin Lispro (Humalog) vs LY900014; <=4 hours post meal; Test type: Other; p = 0.217, Negative binomial regression; Relative rate = 1.22, 95% CI 2-sided [0.89 to 1.68]
Statistical Analysis 5: Comparison: Insulin Lispro (Humalog) vs LY900014; >1 to <=2 hours post meal; Test type: Other; p = 0.703, Negative binomial regression; Relative rate = 1.09, 95% CI 2-sided [0.71 to 1.65]
Statistical Analysis 6: Comparison: Insulin Lispro (Humalog) vs LY900014; >2 to <=4 hours post meal; Test type: Other; p = 0.206, Negative binomial regression; Relative rate = 1.24, 95% CI 2-sided [0.89 to 1.73]
Statistical Analysis 7: Comparison: Insulin Lispro (Humalog) vs LY900014; >4 hours post meal; Test type: Other; p = 0.082, Negative binomial regression; Relative rate = 0.75, 95% CI 2-sided [0.55 to 1.04]

6. Secondary Outcome: Change From Baseline in 1,5-Anhydroglucitol (1,5-AG)
Description: 1,5-anhydroglucitol (1,5-AG) is a marker of short-term glycemic control especially postprandial hyperglycemia. It accurately predicts rapid changes in glycemia and is tightly associated with glucose fluctuations and postprandial glucose. LS mean was determined by MMRM model with Baseline + Pooled Country + Hemoglobin A1c Stratum at Baseline + Use of Metformin at Study Entry + Type of Basal at Lead-in Stratum + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and at least one post-baseline 1,5-AG data.
Measure: Least Squares Mean (Standard Error); unit: milligrams per liter (mg/L)
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 164 | 162
milligrams per liter (mg/L) | 0.39 (0.202) | 0.10 (0.203)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; Test type: Other; p = 0.309, Mixed Models Analysis; LS Mean Difference = -0.29, 95% CI 2-sided [-0.86 to 0.27]

7. Secondary Outcome: Change From Baseline in 10-Point Self-Monitoring Blood Glucose (SMBG) Values
Description: SMBG 10-point profiles were measured at morning (premeal-fasting, 1-hour post meal, 2-hour post meal), midday (premeal, 1-hour post meal, 2-hour post meal), evening (premeal, 1-hour post meal, 2-hour post meal) and bedtime. LS Mean was determined by MMRM model with Baseline + Pooled Country + Hemoglobin A1c Stratum at Baseline + Use of Metformin at Study Entry + Type of Basal at Lead-in Stratum + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and at least one post-baseline SMBG data.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 149 | 149
milligrams per deciliter (mg/dL)
  Morning premeal-fasting | 5.5 (2.90) | -10.2 (2.90)
  Morning 1-hour post meal: number analyzed (Participants) | 147 | 149
  Morning 1-hour post meal | -6.4 (3.53) | -20.4 (3.51)
  Morning 2-hour postmeal: number analyzed (Participants) | 148 | 149
  Morning 2-hour postmeal | -9.5 (3.63) | -24.4 (3.62)
  Midday premeal | -6.7 (3.25) | -9.0 (3.26)
  Midday 1-hour post meal: number analyzed (Participants) | 148 | 149
  Midday 1-hour post meal | -4.7 (3.34) | -13.8 (3.33)
  Midday 2-hour post meal: number analyzed (Participants) | 149 | 148
  Midday 2-hour post meal | -10.8 (3.31) | -14.1 (3.33)
  Evening premeal | -12.2 (4.00) | -1.6 (4.01)
  Evening 1-hour post meal: number analyzed (Participants) | 147 | 149
  Evening 1-hour post meal | -2.4 (3.54) | -8.0 (3.52)
  Evening 2-hour post meal | -7.0 (3.50) | -14.8 (3.50)
  Bedtime: number analyzed (Participants) | 146 | 148
  Bedtime | -7.9 (3.84) | -12.4 (3.82)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; Morning premeal-fasting; Test type: Other; p < .001, Mixed Models Analysis; LS Mean Difference = -15.7, 95% CI 2-sided [-23.8 to -7.7]
Statistical Analysis 2: Comparison: Insulin Lispro (Humalog) vs LY900014; Morning 1-hour post meal; Test type: Other; p = 0.005, Mixed Models Analysis; LS Mean Difference = -14.0, 95% CI 2-sided [-23.8 to -4.2]
Statistical Analysis 3: Comparison: Insulin Lispro (Humalog) vs LY900014; Morning 2-hour post meal; Test type: Other; p = 0.004, Mixed Models Analysis; LS Mean Difference = -14.9, 95% CI 2-sided [-25.0 to -4.8]
Statistical Analysis 4: Comparison: Insulin Lispro (Humalog) vs LY900014; Midday premeal; Test type: Other; p = 0.616, Mixed Models Analysis; LS Mean Difference = -2.3, 95% CI 2-sided [-11.4 to 6.8]
Statistical Analysis 5: Comparison: Insulin Lispro (Humalog) vs LY900014; Midday 1-hour post meal; Test type: Other; p = 0.054, Mixed Models Analysis; LS Mean Difference = -9.1, 95% CI 2-sided [-18.4 to 0.1]
Statistical Analysis 6: Comparison: Insulin Lispro (Humalog) vs LY900014; Midday 2-hour post meal; Test type: Other; p = 0.483, Mixed Models Analysis; LS Mean Difference = -3.3, 95% CI 2-sided [-12.6 to 6.0]
Statistical Analysis 7: Comparison: Insulin Lispro (Humalog) vs LY900014; Evening premeal; Test type: Other; p = 0.064, Mixed Models Analysis; LS Mean Difference = 10.5, 95% CI 2-sided [-0.6 to 21.7]
Statistical Analysis 8: Comparison: Insulin Lispro (Humalog) vs LY900014; Evening 1-hour post meal; Test type: Other; p = 0.262, Mixed Models Analysis; LS Mean Difference = -5.6, 95% CI 2-sided [-15.5 to 4.2]
Statistical Analysis 9: Comparison: Insulin Lispro (Humalog) vs LY900014; Evening 2-hour post meal; Test type: Other; p = 0.117, Mixed Models Analysis; LS Mean Difference = -7.8, 95% CI 2-sided [-17.5 to 2.0]
Statistical Analysis 10: Comparison: Insulin Lispro (Humalog) vs LY900014; Bedtime; Test type: Other; p = 0.414, Mixed Models Analysis; LS Mean Difference = -4.4, 95% CI 2-sided [-15.1 to 6.2]

8. Secondary Outcome: Change From Baseline in Daily Insulin Dose
Description: LS mean was determined by MMRM model with Baseline + Pooled Country + Hemoglobin A1c Stratum at Baseline + Use of Metformin at Study Entry + Type of Basal at Lead-in Stratum + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and at least one post-baseline insulin dose data.
Measure: Least Squares Mean (Standard Error); unit: Units per day
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 168 | 163
Units per day
  Basal Insulin Dose | 0.0 (0.24) | 0.0 (0.24)
  Bolus Insulin Dose | 6.0 (0.69) | 6.6 (0.70)
  Total Insulin Dose | 6.0 (0.75) | 6.6 (0.76)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; Basal insulin dose; Test type: Other; p = 0.947, Mixed Models Analysis; LS Mean Difference = 0.0, 95% CI 2-sided [-0.7 to 0.6]
Statistical Analysis 2: Comparison: Insulin Lispro (Humalog) vs LY900014; Bolus insulin dose; Test type: Other; p = 0.500, Mixed Models Analysis; LS Mean Difference = 0.7, 95% CI 2-sided [-1.3 to 2.6]
Statistical Analysis 3: Comparison: Insulin Lispro (Humalog) vs LY900014; Total insulin dose; Test type: Other; p = 0.543, Mixed Models Analysis; LS Mean Difference = 0.6, 95% CI 2-sided [-1.4 to 2.7]

9. Secondary Outcome: Percentage of Participants With HbA1c <7% and ≤6.5%
Description: HbA1c is the glycosylated fraction of hemoglobin A. It is measured to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: Week 26
Population: All randomized participants with baseline and at least one post-baseline HbA1c data.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 165 | 161
Percentage of participants
  HbA1c < 7% | 28.48 | 26.71
  HbA1c ≤ 6.5% | 15.15 | 9.94
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; For HbA1c < 7%; Test type: Other; p = 0.462, Regression, Logistic; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.47 to 1.42]
Statistical Analysis 2: Comparison: Insulin Lispro (Humalog) vs LY900014; For HbA1c ≤6.5%; Test type: Other; p = 0.089, Regression, Logistic; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.26 to 1.10]

ADVERSE EVENTS:
Time Frame: From baseline until safety follow-up (up to 30 weeks)
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Insulin Lispro (Humalog) | LY900014
All-Cause Mortality (participants affected / at risk) | 0/178 | 0/176
Serious Adverse Events (participants affected / at risk) | 12/178 | 13/176
Other Adverse Events (participants affected / at risk) | 29/178 | 28/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Insulin Lispro (Humalog) (N=178) | LY900014 (N=176)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic complication (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (4)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 1 (1)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1/78 (1) | 1/82 (1)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1/78 (1) | 0/82 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro (Humalog) (N=178) | LY900014 (N=176)
Upper respiratory tract infection (Infections and infestations) | 21 (25) | 21 (25)
Weight increased (Investigations) | 10 (10) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT03952130/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT03952130/SAP_001.pdf